CLINICAL TRIAL: NCT00777296
Title: Phase 2a Multidose Safety and Tolerability Study of Dose Escalation of Liposomal Amikacin for Inhalation (ARIKACE™) In Cystic Fibrosis Patients With Chronic Infections Due To Pseudomonas Aeruginosa.
Brief Title: Multidose Safety and Tolerability Study of Dose Escalation of Liposomal Amikacin for Inhalation (ARIKACE™)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR02-105
Record Dates: First submitted 2008-10-15; First posted 2008-10-22 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Respiratory Infections; Pulmonary Cystic Fibrosis; CFTR
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 - 280 mg ARIKACE™ (Experimental): Subjects in this cohort will receive 280 mg of ARIKACE™
  Interventions: Drug: ARIKACE™
- Cohort 1 - Placebo (Placebo Comparator): Subjects in this arm of cohort 1 will receive matching placebo
  Interventions: Drug: Placebo
- Cohort 2 - 560 mg ARIKACE™ (Experimental): Subjects in this cohort will receive 560 mg of ARIKACE™
  Interventions: Drug: ARIKACE™
- Cohort 2 - Placebo (Placebo Comparator): Subjects in this arm of cohort 2 will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARIKACE™ — Study start date is before Jan 18, 2017.
  Other Names: liposomal amikacin for inhalation; Arikayce
  Arms: Cohort 1 - 280 mg ARIKACE™; Cohort 2 - 560 mg ARIKACE™
Drug: Placebo — Study start date is before Jan 18, 2017.
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo

SUMMARY:
A major factor in the respiratory health of cystic fibrosis (CF) subjects is acquisition of chronic Pseudomonas aeruginosa infections. The infection rate with P. aeruginosa increases with age and by age 18 years, 80% of CF subjects in the U.S. are infected. Liposomal Amikacin for Inhalation (Arikace™) is a sterile aqueous liposomal suspension consisting of amikacin sulfate encapsulated in liposomes. This formulation of amikacin maximizes the achievable dose and delivery to the lungs of subjects infected via a nebulizer. Because liposome particles are small enough to penetrate and diffuse through sputum into the bacterial biofilm, they deposit drug in close proximity to the bacterial colonies, thus improving the bioavailability of amikacin at the infection site. The clinically achievable doses of amikacin in the LAI formulation can effectively increase the half-life of the drug in the lungs, and decrease the potential for systemic toxicity. LAI offers several advantages over current therapies in treating CF subjects with chronic infection caused by P. aeruginosa.

DETAILED DESCRIPTION:
Cystic fibrosis is a genetic disease resulting from mutations in a 230 kb gene on chromosome 7 known as the cystic fibrosis transmembrane conductance regulator (CFTR). Study subjects with CF manifest pathological changes in a variety of organs that express CFTR. The lungs are frequently affected, the sequelae being chronic infections and airway inflammation. The principal goal of treatment of subjects with CF is to slow the chronic deterioration of lung function.

This is a Phase 2a study of safety, and tolerability of 28 days of daily dosing of two dose (280 mg, and 560 mg) cohorts of Arikace™ versus placebo. Study subjects will be randomized to receive either study drug or placebo (1.5% NaCl) by inhalation via a PARI eFlow® nebulizer. Cohort 1 (280mg) will complete 28 days of daily dosing with Arikace™ and 14 day post dosing safety evaluation by the Safety Committee (DSMB) before initiation of enrollment in Cohort 2 (560mg). Cohort 2 will complete 28 days of daily dosing, and a 14 day post dosing safety assessment by the DSMB to evaluate safety data. All study patients will be followed for safety, pharmacokinetics, clinical, and microbiologic activity for 28 days post completion of study treatment.

The total study period will be up to 56 days, with screening visit occurring within the preceding 14 days prior to randomization. Patients will be clinically evaluated during the first 48 hours post-randomization, and weekly for the 28 days treatment period, and during the follow up visits at study days 35, 42, 49, and 56 days to determine safety, tolerability, pharmacokinetics (PK), and clinical, and microbiologic activity.

Clinical laboratory parameters, audiology testing, clinical adverse events, and pulmonary function will be evaluated for all study subjects in order to determine the qualitative and quantitative safety and tolerability of Arikace™ compared to Placebo. Serum, urine, and sputum specimens will be collected at periodic intervals to assess PK. Additionally; sputum samples will be collected to determine changes in bacterial density. Pulmonary function testing and CFQ-R measurements will be assessed at selected time points throughout the study.

DSMB has recommended the amendment of the main study to evaluate safety and efficacy of additional cycles of treatment with Arikace™. All patients who were randomized in the main study, were compliant with the study protocol, and continue meeting study eligibility criteria can be consented to participate in the open-label extension to evaluate the safety, tolerability and efficacy of 560 mg once daily dose of Arikace™ administered for six cycles over eighteen months. Each cycle will comprise of 28 days of treatment followed by 56 days off treatment. The total extension period will be up to 518 days (74 weeks, about 18 months).

Clinical laboratory parameters, audiology testing, clinical adverse events, and pulmonary function will be evaluated for all study subjects in order to determine the longer term safety, tolerability, and efficacy of Arikace™. Serum specimens will be collected at periodic intervals to assess PK for safety. Additionally, sputum samples will be collected to determine changes in bacterial density. Pulmonary function testing and CFQ-R measurements will be assessed at selected time points throughout the study. Arikace™, Arikayce™, Liposomal Amikacin for Inhalation (LAI) and Amikacin Liposome Inhalation Suspension (ALIS) are all the same may be used interchangeably throughout the study and other studies evaluating amikacin liposome inhalation suspension.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from patient or designated legal guardian prior to the performance of any study related procedures.
* Male or female study subjects ≥6 years of age or older
* Confirmed diagnosis of CF
* History of chronic infection with P. aeruginosa
* Study subjects must produce a screening specimen that is positive for growth of P. aeruginosa
* FEV1 ≥ 40% predicted at Screening
* SaO2 ≥ 90% at Screening while breathing room air
* Ability to comply with study medication use, study visits and study procedures as judged by the investigator
* Ability to produce sputum or be willing to undergo an induction to produce sputum for clinical evaluation
* Clinically stable with no evidence of acute upper or lower respiratory tract infection of history of pulmonary exacerbation within 4 weeks prior to screening

Key Exclusion Criteria:

* Administration of any investigational drug within 8 weeks prior to Screening
* Emergency room visit or hospitalization for CF or respiratory-related illness within 4 weeks prior to screening
* History of alcohol, medication or illicit drug abuse within the 1 year prior to screening
* History of lung transplant
* Female of childbearing potential who is lactating or is not practicing an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or IUD)
* Positive pregnancy test
* Use of any anti-pseudomonal anitbiotics (IV antibiotics, all inhalation antibiotics, oral fluoroquinolones)within the 28 days prior to screening
* Initiation of chronic therapy (i.e. TOBI®, high-dose ibuprofen, rhDNase, macrolide antibiotics) within 28 days prior to screening
* History of sputum or throat swab culture yielding Burkholderia cepacia within 2 years of Screening
* History of mycobacterial or Aspergillus infection
* Requiring treatment within 2 years prior to screening, and/or history of allergic bronchopulmonary aspergillosis.
* History of biliary cirrhosis with portal hypertension, or splenomegaly
* History of daily, continuous oxygen supplementation or requirement for more than 2 L/min at night Change in chest x-ray at screening (or within the 3 months prior to screening)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-02-22 (Actual); Primary Completion 2008-02-27 (Actual); Study Completion 2008-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated
Locations (11):
- Leuven, Belgium
- Hungary (2):
  - Budapest
  - Kaposvár
- Skopje, North Macedonia
- Poland (2):
  - Rabka-Zdrój
  - Warsaw
- Belgrade, Serbia
- Slovakia (2):
  - Bratislava
  - Košice
- Ukraine (2):
  - Kharkiv
  - Kiev

REFERENCES:
- [Background] Clancy JP, Dupont L, Konstan MW, Billings J, Fustik S, Goss CH, Lymp J, Minic P, Quittner AL, Rubenstein RC, Young KR, Saiman L, Burns JL, Govan JR, Ramsey B, Gupta R; Arikace Study Group. Phase II studies of nebulised Arikace in CF patients with Pseudomonas aeruginosa infection. Thorax. 2013 Sep;68(9):818-25. doi: 10.1136/thoraxjnl-2012-202230. Epub 2013 Jun 8. PMID 23749840
- [Background] Okusanya OO, Bhavnani SM, Hammel JP, Forrest A, Bulik CC, Ambrose PG, Gupta R. Evaluation of the pharmacokinetics and pharmacodynamics of liposomal amikacin for inhalation in cystic fibrosis patients with chronic pseudomonal infections using data from two phase 2 clinical studies. Antimicrob Agents Chemother. 2014 Sep;58(9):5005-15. doi: 10.1128/AAC.02421-13. Epub 2014 Mar 31. PMID 24687506
- [Background] Meers P, Neville M, Malinin V, Scotto AW, Sardaryan G, Kurumunda R, Mackinson C, James G, Fisher S, Perkins WR. Biofilm penetration, triggered release and in vivo activity of inhaled liposomal amikacin in chronic Pseudomonas aeruginosa lung infections. J Antimicrob Chemother. 2008 Apr;61(4):859-68. doi: 10.1093/jac/dkn059. Epub 2008 Feb 27. PMID 18305202

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - 280 mg ARIKACE™: Subjects in this cohort received 280 mg of ARIKACE™
- Cohort 1 - Placebo: Subjects in this arm of cohort 1 received matching placebo
- Cohort 2 - 560 mg ARIKACE™: Subjects in this cohort received 560 mg of ARIKACE™
- Cohort 2 - Placebo: Subjects in this arm of cohort 2 received matching placebo
Period: Overall Study
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 1 - Placebo | Cohort 2 - 560 mg ARIKACE™ | Cohort 2 - Placebo
Started | 21 | 11 | 23 | 11
Completed | 20 | 10 | 21 | 10
Not Completed | 1 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — CRF form not completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 1 - Placebo | Cohort 2 - 560 mg ARIKACE™ | Cohort 2 - Placebo | Total
Number analyzed (Participants) | 21 | 11 | 23 | 11 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (5.3) | 16.9 (7.9) | 16.6 (6.1) | 17.2 (5.8) | 16.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 11 | 4 | 39
  Male | 5 | 3 | 12 | 7 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian (not of Hispanic origin) | 21 | 11 | 23 | 11 | 66

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Laboratory Abnormalities.
Description: Changes in chemistry and hematology lab tests (clinically significant value of CTCAE grade ≥ 3).
Time Frame: 28 Days
Population: The analysis population is the modified intent-to-treat (mITT) population, defined as all randomized subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - Placebo: Subjects in this cohort who received placebo
- Cohort 2 - Placebo: Subjects in this cohort received matching placebo
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 1 - Placebo | Cohort 2 - 560 mg ARIKACE™ | Cohort 2 - Placebo
Number analyzed (Participants) | 21 | 11 | 21 | 11
Participants
  Neutrophils absolute | 1 | 0 | 8 | 7
  Leucocytes | 1 | 0 | 3 | 3
  Glucose | 0 | 0 | 2 | 0
  Lymphocytes absolute | 1 | 0 | 2 | 0
  Calcium | 0 | 0 | 1 | 0
  Creatinine clearance | 0 | 0 | 1 | 0
  Potassium | 3 | 1 | 1 | 0

2. Secondary Outcome: Pharmacokinetics (PK) of Arikace™ in Serum.
Description: Measure PK parameters (AUC0-infinity) of Arikace™ in serum.
Time Frame: Day 1, Day 14 and Day 28
Population: The PK population consisted of subjects who received amikacin, had at least one serum PK assessment and were not replaced.
Measure: Mean (Standard Deviation); unit: mg.hr/L
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 2 - 560 mg ARIKACE™
Number analyzed (Participants) | 21 | 21
mg.hr/L
  Day 1 | 5.73 (3.40) | 7.92 (3.55)
  Day 14 | 7.61 (4.04) | 12.5 (10.9)
  Day 28 | 8.03 (6.12) | 14.6 (11.7)

3. Secondary Outcome: Pharmacokinetic (PK) of Arikace in Serum (Cmax).
Description: Measure PK parameter (Cmax) of Arikace™ in serum.
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 2 - 560 mg ARIKACE™
Number analyzed (Participants) | 21 | 21
mg/L
  Day 1 | 0.95 (0.58) | 1.08 (0.51)
  Day 14: number analyzed (Participants) | 20 | 21
  Day 14 | 1.28 (1.02) | 1.84 (1.35)
  Day 28: number analyzed (Participants) | 20 | 21
  Day 28 | 1.42 (1.45) | 2.27 (1.58)

4. Secondary Outcome: Pharmacokinetics (PK) of Arikace™ in Sputum (AUC).
Description: Measure PK parameter (AUC0-24) of Arikace™ in sputum.
Time Frame: 28 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg*hr/g
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 2 - 560 mg ARIKACE™
Number analyzed (Participants) | 21 | 21
mcg*hr/g | 13120 (21386) | 22445 (18652)

5. Secondary Outcome: Pharmacokinetics (PK) of Arikace™ in Urine.
Description: Measure PK parameter (Ae0-24 (mg) of Arikace™.
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 2 - 560 mg ARIKACE™
Number analyzed (Participants) | 21 | 21
mg
  Day 1: number analyzed (Participants) | 21 | 20
  Day 1 | 17.7 (12.3) | 27.0 (25.2)
  Day 14: number analyzed (Participants) | 19 | 20
  Day 14 | 27.3 (16.5) | 39.8 (42.7)
  Day 28: number analyzed (Participants) | 20 | 21
  Day 28 | 25.2 (19.5) | 43.7 (48.9)

6. Secondary Outcome: Sputum Amikacin Levels of Arikace™.
Description: Measure PK parameter (sputum amicakin concentration) of Arikace™ in sputum.
Time Frame: Day 1, Day 14 and Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/g
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 2 - 560 mg ARIKACE™
Number analyzed (Participants) | 21 | 21
mcg/g
  Day 1 | 1197 (1.56) | 2395 (0.866)
  Day 14 | 1174 (1.01) | 3496 (0.973)
  Day 28 | 1911 (1.28) | 2635 (1.23)

7. Secondary Outcome: Pulmonary Function: FEV1 %-Predicted.
Description: Relative Change (%) from Baseline to End of treatment (Day 28) and Day 56 in Pulmonary Function.
Time Frame: Baseline, Day 28, and Day 56
Population: The analysis population is the modified intent-to-treat (mITT) population, defined as all randomized subjects who received at least one dose of study drug.
  Placebo is a pooled value from cohort 280 mg and cohort 560 mg.
Measure: Mean (Standard Deviation); unit: Relative Percent (%) change in FEV1
Groups:
- 280 mg ARIKACE™: Subjects in this cohort received 280 mg of ARIKACE™
- 560 mg ARIKACE™: Subjects in this cohort received 560 mg of ARIKACE™
- Pooled Placebo: Subjects in this arm received matching placebo
Arm/Group | 280 mg ARIKACE™ | 560 mg ARIKACE™ | Pooled Placebo
Number analyzed (Participants) | 21 | 21 | 22
Relative Percent (%) change in FEV1
  Baseline | 66.4 (20.0) | 62.9 (18.2) | 68.0 (22.4)
  Day 28 | 9.6 (13.7) | 11.0 (16.4) | 0.5 (10.5)
  Day 56 | 1.8 (8.8) | 13.8 (26.2) | -3.8 (13.5)

8. Secondary Outcome: Pulmonary Function: FEV1.
Description: Mean Percent Change (%) from Baseline to End of treatment (Day 28) and Day 56 in Pulmonary Function.
Time Frame: Baseline, Day 28, and Day 56
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Mean Percent (%) Change in FEV1
Arm/Group | 280 mg ARIKACE™ | 560 mg ARIKACE™ | Pooled Placebo
Number analyzed (Participants) | 21 | 21 | 22
Mean Percent (%) Change in FEV1
  Baseline | 2.022 (0.788) | 1.937 (0.936) | 1.968 (0.654)
  Day 28 | 10.1 (12.8) | 13.2 (16.2) | 2.2 (11.9)
  Day 56 | 2.0 (8.6) | 13.2 (24.3) | -4.4 (13.0)

9. Secondary Outcome: Change From Baseline in Log10CFU Per Gram (Density) of Pseudomonas Aeruginosa in Sputum.
Description: End-of-treatment (Day 28) from baseline in density of P. aeruginosa (log10 CFU/g) in sputum.
Time Frame: Day 7, Day 14, Day 21, Day 28 and Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10CFU per gram
Arm/Group | 280 mg ARIKACE™ | 560 mg ARIKACE™ | Pooled Placebo
Number analyzed (Participants) | 21 | 21 | 22
log10CFU per gram
  Day 7 | 0.080 (1.882) | -1.101 (2.170) | 0.052 (1.303)
  Day 14 | -1.366 (2.013) | -1.570 (2.161) | -0.574 (1.006)
  Day 21 | -1.044 (2.155) | -2.283 (2.775) | -0.440 (1.280)
  Day 28 | -0.622 (1.881) | -1.515 (1.699) | -0.677 (1.043)
  Day 35 | -0.380 (1.425) | -1.313 (2.852) | -0.445 (1.201)

10. Secondary Outcome: Duration of Systemic Antipseudomonal Rescue Therapy.
Description: Duration of systemic antipseudomonal rescue therapy during the study in both the ARIKACE™ and placebo groups.
Time Frame: Through study duration, approximately 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Groups:
- ARIKACE™ 280 mg: Subjects who received the 280 mg dose of the ARIKACE™
- Placebo for ARIKACE™ 280 mg: Subjects who received matching placebo for ARIKACE™ 280 mg dose.
- ARIKACE™ 560 mg: Subjects who received the 560 mg dose of the ARIKACE™
- Placebo for ARIKACE™ 560 mg: Subjects who received matching placebo for ARIKACE™ 560 mg dose.
Arm/Group | ARIKACE™ 280 mg | Placebo for ARIKACE™ 280 mg | ARIKACE™ 560 mg | Placebo for ARIKACE™ 560 mg
Number analyzed (Participants) | 21 | 11 | 21 | 11
days | 14.00 (0.00) | 27.00 (NA) — Standard deviation does not apply because only 1 participant required rescue therapy | 19.00 (NA) — Standard deviation does not apply because only 1 participant required rescue therapy | 21.00 (11.31)

11. Secondary Outcome: Number of Subjects Requiring Antipseudomonal Rescue Therapy.
Description: Number of Subjects requiring systemic antipseudomonal rescue therapy during the study in both the ARIKACE™ and placebo groups.
Time Frame: Through study duration, approximately 56 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- ARIKACE™: Subjects who received either the 280 mg or the 560 mg doses of the ARIKACE™
- Placebo: Subjects who received matching placebo.
Arm/Group | ARIKACE™ | Placebo
Number analyzed (Participants) | 42 | 22
Participants | 4 | 3

12. Secondary Outcome: CFQ-R Respiratory Scale (Absolute Change From Baseline).
Description: Quality of Life was measured by the absolute change from baseline in the Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory scale. Disease specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms in patients with a diagnosis of cystic fibrosis. Scores range from 0 to 100, with higher scores indicating better health. Scores for each Health Related Quality of Life (HRQoL) domain; after recoding, each item is summed to generate a domain score and standardized.
Time Frame: Baseline/Day 1, Day 15, Day 28 and Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 1 - Placebo | Cohort 2 - 560 mg ARIKACE™ | Cohort 2 - Placebo
Number analyzed (Participants) | 21 | 11 | 21 | 11
score on a scale
  Day 1/baseline | 72.619 (11.630) | 71.212 (14.921) | 67.989 (12.748) | 61.364 (21.425)
  Day 15 | 2.632 (10.078) | -0.505 (12.349) | 3.704 (16.133) | -2.778 (16.054)
  Day 28 | 4.306 (12.760) | -3.283 (14.154) | 5.688 (11.669) | 1.667 (13.302)
  Day 42 | 1.080 (12.169) | -4.012 (19.598) | 3.042 (18.213) | 0.556 (12.200)

ADVERSE EVENTS:
Time Frame: AEs were assessed from the first dose (Visit 2) until the completion of the study follow-up (14 days after 28 days of dosing in cohort 2). The total duration is approximately 84 days.
Arm/Group | Cohort 1 - 280 mg ARIKACE™ | Cohort 1 - Placebo | Cohort 2 - 560 mg ARIKACE™ | Cohort 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11 | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/11 | 2/21 | 1/11
Other Adverse Events (participants affected / at risk) | 10/21 | 6/11 | 5/21 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 280 mg ARIKACE™ (N=21) | Cohort 1 - Placebo (N=11) | Cohort 2 - 560 mg ARIKACE™ (N=21) | Cohort 2 - Placebo (N=11)
ENTEROVIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 280 mg ARIKACE™ (N=21) | Cohort 1 - Placebo (N=11) | Cohort 2 - 560 mg ARIKACE™ (N=21) | Cohort 2 - Placebo (N=11)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
PHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other